CLINICAL TRIAL: NCT01856452
Title: Phase II Study of Comparison of Sentinel Lymph Node Biopsy Guided by The Multimodal Method of Indocyanine Green Fluorescence, Radioisotope and Blue Dye Versus the Radioisotope in Breast Cancer
Brief Title: Comparison Study of Sentinel Lymph Node Biopsy by Multimodal Method in Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, So-Youn Jung, Medical Doctor, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCC-1110212-2
Record Dates: First submitted 2013-05-08; First posted 2013-05-17 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Breast Neoplasms
Keywords: Sentinel lymph node; multimodal; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- radioisotope (Active Comparator): sentinel lymph node operation using radioisotope in the breast cancer patients
  Interventions: Device: radioisotope
- the mixture including indocyanine green (Experimental): sentinel lymph node operation using the mixture of indocyanine green, blue dye and radioisotope in the breast cancer patients
  Interventions: Device: the mixture including indocyanine green

INTERVENTIONS:
Device: the mixture including indocyanine green — Sentinel lymph node biopsy using near-infrared imaging system and gamma probe detector for the mixture of indocyanine green, blue dye, and radioisotope during operation
  Arms: the mixture including indocyanine green
Device: radioisotope — Sentinel lymph node biopsy using gamma probe detector for radioisotope during operation
  Arms: radioisotope

SUMMARY:
Sentinel lymph node biopsy (SLNB) has become a mainstay surgery method in breast cancer. It provides the surgeon the evidence of axillary lymph node metastasis, which determines the extent of surgery. Because effective SLNB can decrease the extent of axillary lymph node dissection, it is increasingly important. In general, radioactive colloid has been used for SLNB. In order to pursue more precise SLNB, the investigators developed a multimodal method enabling visual guidance with the mixture of indocyanine green, blue dye and radioisotope.

In this study, our hypotheses are as following:

1. Multimodal method enables to increase identification rate of SLNB
2. blue dye and indocyanine green provide the surgeon visual guidance to ensure better outcome
3. Multimodal method alleviates the shortcomings of indocyanine green and blue dye as an identification strategy

DETAILED DESCRIPTION:
Indocyanine green Advantages: provides visualization of sentinel lymph node without incision

Blue dye Advantages: easy to employ; no toxicity Disadvantages: diffusion; absorption and disappearance of the marking within minutes

Radioisotope Advantages: can be used for lesions not accessible to Ultrasound; ideal for selective uptake to sentinel lymph node Disadvantages: not able to use palpation and visualization, confirms by gamma-probe only

ELIGIBILITY:
Inclusion Criteria:

* clinically lymph node negative breast cancer patients
* consented patients with more than 20 years

Exclusion Criteria:

* history of breast cancer
* locally advanced breast cancer and metastatic breast cancer
* proven axillary lymph node metastasis
* history of axillary excisional or incisional biopsy, or dissection
* history of neoadjuvant chemotherapy
* pregnancy
* non-consented patients
* younger than 20 years old

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Time to sentinel lymph node biopsy | up to 6 months
  From the date of randomization, skin necrosis and dye staining are assessed up to 6 months after the operation (post op 3 mon and 6 mon follow-up).

SECONDARY OUTCOMES:
Identification rate of sentinel lymph node biopsy | 13 months
  The number of participants with sentinel lymph node detection is assessed up to 13 months.

CONTACTS AND LOCATIONS:
Overall Officials: So-Youn Jung, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea